CLINICAL TRIAL: NCT00836108
Title: Unsupported Arm Exercise and Breathing Strategy in Patients With Chronic
Brief Title: Unsupported Arm Exercise and Breathing Strategy in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Directory Respiratory Medicine, West Park Healthcare Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RG20080707ArmStrategy
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Lung Diseases, Obstructive; Breathing Exercises; Exercise Tolerance; Dyspnea; Arm Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Sham Comparator): spontaneous
  Interventions: Behavioral: breathing strategy
- 2 (Experimental): coordinating arm elevation with inspiration
  Interventions: Behavioral: breathing strategy
- 3 (Experimental): coordinating arm elevation with expiration
  Interventions: Behavioral: breathing strategy

INTERVENTIONS:
Behavioral: breathing strategy — Subjects will practice a rhythmic overhead arm exercise, during which they will be taught to inspire when they elevate their arms or they will be taught to expire when they elevate their arms or, a third group, will practice a rhythmic overhead arm exercise, during which they will not be provided with any instruction regarding a specific breathing pattern. The arm exercise practiced by all groups will be identical.

SUMMARY:
Controlling the way people with lung problems breathe during arm exercises may reduce their breathlessness during activities of daily living that require them to lift their arms (i.e. brushing their hair, putting groceries away on high shelves). The main aim of this study is to determine the effects of specific breathing strategies during arm exercise on dyspnoea in patients with chronic lung disease. Coordinating inspiration with the action of arm elevation will reduce dyspnoea during a rhythmic overhead arm activity

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD including forced expiratory volume in one second < 80% predicted normal
* presence of lung hyperinflation at rest

Exclusion Criteria:

* musculoskeletal or neurological condition which could adversely affect arm activity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Dyspnoea during arm exercise | 1 week

SECONDARY OUTCOMES:
Arm exercise endurance | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Dina Brooks, PhD, Principal Investigator — West Park Healthcare Centre
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dolmage TE, Janaudis-Ferreira T, Hill K, Price S, Brooks D, Goldstein RS. Arm elevation and coordinated breathing strategies in patients with COPD. Chest. 2013 Jul;144(1):128-135. doi: 10.1378/chest.12-2467. PMID 23370697